CLINICAL TRIAL: NCT03777995
Title: Reliability and Validity of a New Designed Balance Platform for Children
Brief Title: A New Designed Balance Platform for Children
Status: Completed | Type: Observational
Sponsor: Eastern Mediterranean University (Other)
Responsible Party: Sponsor
Other Study IDs: ETK00-2018-0204
Record Dates: First submitted 2018-12-14; First posted 2018-12-19 (Actual); Last update posted 2019-10-24 (Actual); Status verified 2018-12

CONDITIONS: Child Development
Keywords: Balance

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
People always come across with different floors which gradually affect dynamic balance. Dynamic balance is important in activities of daily life of all people. There are various reliable and valid tests for both children and adults, but no test design which includes different floor materials has been developed. Thus, this study aimed to describe a new designed balance test platform and investigate its reliability and validity in 3-5 years old children.

DETAILED DESCRIPTION:
Children whose families signed consent form will be included. Height and weight will be measured. Then they will be taken to the balance measurements. Design will firstly be shown to child and one trial will be permitted before starting the test. Timed-up and Go test will also be used as a reliable and valid test for dynamic balance in this age group. Single leg standing will also be used to investigate the discrimination feature of the dynamic balance tested by new design platform.

All tests will be done without socks and shoes. Timing will be the only results for all tests. Calibrated chronometers will be used for this aim. After all measurements complete, statistical analysis will be conducted.

ELIGIBILITY:
Inclusion Criteria:

* Chid aged 3-5 years (birth date: December 2013 - December 2015)
* Parents who signed consent form.

Exclusion Criteria:

* Children who have problem about musculoskeletal system, neurological disorder, vestibular system disorders.
* Children who mention painful situations which may possibly prevent to walk on the platform
* Children who have visual problems

Ages: 3 Years to 5 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Children who have a typical development will be recruited from various kindergartens in Cyprus.
Sampling Method: Probability Sample
Enrollment: 108 (Actual)
Dates: Start 2018-12-15 (Actual); Primary Completion 2019-03-10 (Actual); Study Completion 2019-04-10 (Actual)

PRIMARY OUTCOMES:
New designed test | at baseline
  This is a walking platform which has different floor materials

SECONDARY OUTCOMES:
Timed-up and go test | at baseline
  This is a reliable and valid test which is used to assess dynamic balance in children. There is a three meter pathway. Two chairs are used for the starting point and to specify the returning point. The test will be repeated 3 times and the best completion time will be recorded.
Single leg standing | at baseline
  Children are asked to stand on dominant leg. Their standing duration will be recorded.

CONTACTS AND LOCATIONS:
Overall Officials: ZEHRA GÜÇHAN TOPCU, Principal Investigator — Eastern Mediterranean University
Locations (1):
- Zehra Güçhan Topcu, Famagusta, Cyprus